CLINICAL TRIAL: NCT03891121
Title: Which One is Effective in Treatment of Bruxism? Occlusal Splints or Botulinum Toxin
Brief Title: Occlusal Splints or Botulinum Toxin?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Mehmet Emre Yurttutan, DDS, PhD, Oral and Maxillofacial Surgery Specialist, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36290600/49
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Myofascial Pain; Temporomandibular Disorder
Keywords: Myofascial Pain; Botulinum Toxin
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Occlusal Splints; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Occlusal splint (Experimental): Patients were treated with occlusal splint.
  Interventions: Device: Occlusal Splint
- Botulinum toxin (Experimental): Patients were treated with botulinum toxin injection.
  Interventions: Drug: Botulinum toxin type A
- Both (Experimental): Patients were treated with occlusal splint and botulinum toxin injection together.
  Interventions: Device: Occlusal Splint; Drug: Botulinum toxin type A

INTERVENTIONS:
Device: Occlusal Splint — Occlusal splints are appliances that were usually applied to the upper jaw and covering all teeth and they are made of autopolymerizing acrylic resin. It is produced by using 2 mm thick hard acrylic between the maxilla and mandible as defined by the Okeson.
  Arms: Both; Occlusal splint
Drug: Botulinum toxin type A — We diluted 100-U freeze-dried BTX-A with 1.0 milliliters of sodium chloride, resulting in a dose of 1.0 U per 0.1 mL. We administered all skin injections by using a 1-inch 30-gauge needle. Patients were placed with the Frankfurt horizontal plane parallel to the floor.
  Arms: Both; Botulinum toxin

SUMMARY:
73 patients with myofascial pain due to bruxism were included in this study. The patient were allocated into three groups. Group A was treated with occlusal splint, Group B was treated with botulinum toxin injection, Group C was treated with occlusal splint and botulinum toxin injection together. Temporomandibular Disorder Pain Screener (TMD-PS), Graded Chronic Pain Scale (GCPS), Oral Behavior Checklist (OBC), Jaw Function Limitation Scale (JFLS), Visual Analog Scale (VAS) by palpation of the chewing muscles were administered to all patients before treatment and at 6 months after treatment.

DETAILED DESCRIPTION:
A number of 173 patients were examined for myofascial pain due to TMD in the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Ankara University between April-August 2018. An informed consent was taken from all the patients after obtaining Institutional Ethical Committee approval. The study was performed in accordance with the Helsinki Declaration and all participants signed an informed consent agreement. Patients were included in this randomized, blinded, prospective study accordance with the Consolidated Standards of Reporting Trials (CONSORT) statement and the study was performed by blinded three examiners.

Patients older than 18 years with chronic myofascial pain, more than 6 months with myofascial pain, diagnosis of myofascial pain according to the Research Diagnostic Criteria (RDC) of TMD were included to the study. Patients having intracapsular TMD (disc displacement with or without reduction), a history of any treatment for bruxism, patients taking aminoglycosides, penicillamine, quinine and calcium blockers, pregnant or lactating mothers, having neuromuscular disorder (e.g. Orofacial tardive dyskinesia, Lambert-Eaton Syndrome, Myasthenia gravis), having rheumatoid arthritis, having temporomandibular joint osteoarthrosis with radiographic signs, history of previous joint surgery, patients who had undergone botulinum toxin (BTX) treatment before or an allergy to BTX-A were excluded from the study.

The patients who have myofascial pain were diagnosed and examined with using RDC/TMD diagnostic categories I in the RDC/ TMD by first examiner (M.E.Y) and 102 patients fulfilled inclusion criteria. 8 patients did not agree to participate. 94 patients were allocated to 3 groups according to a computer-generated randomization code. Block randomization was done. Patient groups were as follows:

Group A was treated with occlusal splint Group B was treated with botulinum toxin injection, Group C was treated with occlusal splint and botulinum toxin injection together Visual Analog Scale (VAS), TMD Pain Screener(TMD-PS), Graded Chronic Pain Scale (GCPS), Oral Behavior Checklist (OBC), Jaw Function Limitation Scale (JFLS) were administered to all patients before treatment and at 6th months after treatment by third examiner (K.T.S). Patients' pain was examined by palpation of the chewing muscles and the pain was marked from 0 to 10 on the VAS before and after the treatment.

Questionnaires TMD Pain Screener is a self-report, simple, reliable questionnaire used to assess for the presence of any pain-related TMD. Full version with 6 questions were applied. The total score is between 0 and 7. If the total score is between 0 and 3 points, there is no TMD. If the total score is between 4 and 7, there is TMD.

Graded Chronic Pain Scale is a reliable, short and valid tool that evaluates pain intensity and pain related disability with 7 questions. After the scoring, it is classified to 5 grades. Grade 0 with no intensity and disability, Grade 1 with low intensity and low disability, Grade 2 high intensity and low disability, Grade 3 with high disability and moderately limiting, Grade 4 with high disability and severely limiting.

Jaw Function Limitation Scale evaluates the universal limitations on chewing, jaw mobility, verbal and emotional expression. The patient indicates the level of limitation the mentioned activities from 0 to 10.

Oral Behaviors Checklist evaluates the effects of oral parafunctional habits on the masticatory system and the frequency of these habits. Scoring can be computed as the sum of the number of 21 items and the total score is between 21 and 105.

Occlusal splint therapy Occlusal splints are appliances that were usually applied to the upper jaw and covering all teeth and they are made of autopolymerizing acrylic resin. It is produced by using 2 mm thick hard acrylic between the maxilla and mandible as defined by the Okeson. In the centric relationship the buccal cusp tips and incisal edges should be in contact at the same time, there should be canine protection during eccentric movements. The patients were instructed to wear the occlusal splints 12 h/d for 6 months. Patients were called back for follow-up visits at 7th day, 3rd and 6th months after splint insertion. When necessary, additional adjustments were performed.

Injection technique Patients were informed of the possible side effects of botulinum toxin injections and informed consent was obtained from each patient before starting the procedure.

We diluted 100-U freeze-dried BTX-A (Botox, Allergan, Inc., Irvine, CA) with 1.0 milliliters of sodium chloride, resulting in a dose of 1.0 U per 0.1 mL. We administered all skin injections by using a 1-inch 30-gauge needle. Patients were placed with the Frankfurt horizontal plane parallel to the floor.

Skin areas were cleaned and dried with povidone iodine. 5 points for masseter and 3 points for temporalis were marked. The posterior, upper and lower limits of the masseter were determined for safe injection before injection. Before the injection, the patient was instructed to clench the teeth to make injection sites more prominent and the muscles were determined. The needle was placed perpendicular to the skin. After the aspiration, injections were gradually applied to minimize the spread of BTX-A to adjacent anatomical areas. . Second examiner (A.M.T) administered all injections throughout the study. All injections were performed by the same maxillofacial surgeon 90 U of BTX-A in each participant were performed, 15 U into each temporalis muscle, and 30 U into each masseter muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with chronic myofascial pain
* More than 6 months with myofascial pain
* Diagnosis of myofascial pain according to the RDC/TMD

Exclusion Criteria:

* Patients having intracapsular TMD (disc displacement with or without reduction)
* A history of any treatment for bruxism, patients taking aminoglycosides
* Penicillamine
* Quinine and calcium blockers
* Pregnant or lactating mothers
* Having neuromuscular disorder (e.g. Orofacial tardive dyskinesia, Lambert-Eaton Syndrome, Myasthenia gravis)
* Having rheumatoid arthritis
* Having temporomandibular joint osteoarthrosis with radiographic signs
* History of previous joint surgery
* Patients who had undergone BTX treatment before or an allergy to BTX-A

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
VAS | 1 minute
  Visual Analog Scale:Patients' pain was examined by palpation of the chewing muscles and the pain was marked from 0 to 10 on the VAS before and after the treatment. Higher values represent a worse outcome.
TMD-PS | 2 minutes
  TMD Pain Screener is a self-report, simple, reliable questionnaire used to assess for the presence of any pain-related TMD. Full version with 6 questions were applied. The total score is between 0 and 7. If the total score is between 0 and 3 points, there is no TMD. If the total score is between 4 and 7, there is TMD. Higher values represent a worse outcome.
GCPS | 2 minutes
  Graded Chronic Pain Scale is a reliable, short and valid tool that evaluates pain intensity and pain related disability with 7 questions. After the scoring, it is classified to 5 grades. Grade 0 with no intensity and disability, Grade 1 with low intensity and low disability, Grade 2 high intensity and low disability, Grade 3 with high disability and moderately limiting, Grade 4 with high disability and severely limiting. Higher values represent a worse outcome.
JFLS | 3 minutes
  Jaw Function Limitation Scale evaluates the universal limitations on chewing, jaw mobility, verbal and emotional expression. The patient indicates the level of limitation the mentioned activities from 0 to 10.Higher values represent a worse outcome.
OBC | 5 minutes
  Oral Behaviors Checklist evaluates the effects of oral parafunctional habits on the masticatory system and the frequency of these habits. Scoring can be computed as the sum of the number of 21 items and the total score is between 21 and 105. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohrbach R, Larsson P, List T. The jaw functional limitation scale: development, reliability, and validity of 8-item and 20-item versions. J Orofac Pain. 2008 Summer;22(3):219-30. PMID 18780535
- [Background] Freund B, Schwartz M, Symington JM. Botulinum toxin: new treatment for temporomandibular disorders. Br J Oral Maxillofac Surg. 2000 Oct;38(5):466-71. doi: 10.1054/bjom.1999.0238. PMID 11010775
- [Background] Lee SJ, McCall WD Jr, Kim YK, Chung SC, Chung JW. Effect of botulinum toxin injection on nocturnal bruxism: a randomized controlled trial. Am J Phys Med Rehabil. 2010 Jan;89(1):16-23. doi: 10.1097/PHM.0b013e3181bc0c78. PMID 19855255
- [Result] Guarda-Nardini L, Manfredini D, Salamone M, Salmaso L, Tonello S, Ferronato G. Efficacy of botulinum toxin in treating myofascial pain in bruxers: a controlled placebo pilot study. Cranio. 2008 Apr;26(2):126-35. doi: 10.1179/crn.2008.017. PMID 18468272
- [Result] Kurtoglu C, Gur OH, Kurkcu M, Sertdemir Y, Guler-Uysal F, Uysal H. Effect of botulinum toxin-A in myofascial pain patients with or without functional disc displacement. J Oral Maxillofac Surg. 2008 Aug;66(8):1644-51. doi: 10.1016/j.joms.2008.03.008. PMID 18634953